CLINICAL TRIAL: NCT04053270
Title: A Phase III, Multicentre, Randomised, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Subcutanenous Bioresorbable CUV1647 Implants in Patients With Erythropoietic Protoporphyria (EPP)
Brief Title: Multicentre Phase III Erythropoietic Protoporphyria Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUV017
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Erythropoietic Protoporphyria
Keywords: Erythropoietic Protoporphyria; EPP; Afamelanotide
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — afamelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A was administered active implants on Days 0, 120, 240 and placebo implants on Days 60, 180, 300
  Interventions: Drug: Afamelanotide; Drug: Placebo
- Group B (Placebo Comparator): Group B was administered placebo implants on Days 0, 120, 240 and active implants on Days 60, 180, 300
  Interventions: Drug: Afamelanotide; Drug: Placebo

INTERVENTIONS:
Drug: Afamelanotide — 16mg subcutaneous implant
Drug: Placebo — Placebo subcutaneous implant

SUMMARY:
This was a phase III, multicentre, randomised, double-blind, placebo-controlled study, to evaluate the safety and efficacy of subcutaneous bioresorbable afamelanotide implants in patients with Erythropoietic Protoporphyria (EPP).

The study was conducted with two parallel study arms with crossover between treatments every 60 days.

Eligible patients were randomised to a treatment group, and received implants of active treatment (afamelanotide 16mg) or placebo, in an alternating crossover fashion according to the following dosing regime:

* Group A was administered active implants on Days 0, 120, 240 and placebo implants on Days 60, 180, 300
* Group B was administered placebo implants on Days 0, 120, 240 and active implants on Days 60, 180, 300

DETAILED DESCRIPTION:
Afamelanotide is a man-made drug being studied for use as a preventative medication for Erythropoietic Protoporphyria (EPP) sufferers. It is a synthetically produced analogue of human alpha melanocyte stimulating hormone (alpha-MSH).

The study will involve the use of an implant, which comes in the form of a small rod to be administered under the skin. The implant may contain the study drug afamelanotide or a placebo (inactive medication).

This study aims to provide insight into the effectiveness of afamelanotide under normal conditions of use in EPP patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a diagnosis of EPP (confirmed by elevated free protoporphyrin in peripheral erythrocytes) of sufficient severity that they have requested treatment to alleviate their symptoms.
* Aged 18-70 years.
* Written informed consent prior to the performance of any study-specific procedure.

Exclusion Criteria:

* Any allergy to afamelanotide or the polymer contained in the implant or to lignocaine or other local anaesthetic used during the administration of study medication.
* EPP patients with significant hepatic involvement.
* Personal history of melanoma or dysplastic nevus syndrome.
* Current Bowen's disease, basal cell carcinoma, squamous cell carcinoma, or other malignant or premalignant skin lesions.
* Any other photodermatosis such as PLE, DLE or solar urticaria.
* Diagnosed with HIV/AIDS or hepatitis.
* Any evidence of clinically significant organ dysfunction or any clinically significant deviation from normal in the clinical or laboratory determinations.
* Acute history of drug or alcohol abuse (in the last 12 months).
* History of disorders of the gastrointestinal, hepatic, renal, cardiovascular, respiratory, endocrine (including diabetes, Cushing's syndrome, Addison's disease, Peutz-Jeagher syndrome), neurological (including seizures), haematological (especially anaemia of less than 10 g/100 mL) or systemic disease judged to be clinically significant by the Investigator.
* Major medical or psychiatric illness
* Patient assessed as not suitable for the study in the opinion of the investigator (e.g. noncompliance history allergic to local anaesthetics, faints when given injections or giving blood).
* Female who was pregnant (confirmed by positive serum β-HCG pregnancy test prior to baseline) or lactating.
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device).
* Participation in a clinical trial of an investigational agent within 30 days prior to the screening visit.
* Use of regular medications as specified in protocol Section 5.4 Prior and Concomitant Therapy.
* Any factors that may affect skin reflectance measurements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2009-12-09 (Actual); Study Completion 2009-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Development, Study Director — CLINUVEL PHARMACEUTICALS LTD

REFERENCES:
- [Result] Dwyer T, Muller HK, Blizzard L, Ashbolt R, Phillips G. The use of spectrophotometry to estimate melanin density in Caucasians. Cancer Epidemiol Biomarkers Prev. 1998 Mar;7(3):203-6. PMID 9521433

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Group A was administered active implants on Days 0, 120, 240 and placebo implants on Days 60, 180, 300.
  Afamelanotide: 16mg subcutaneous implant Placebo: Placebo subcutaneous implant
- Group B: Group B was administered placebo implants on Days 0, 120, 240 and active implants on Days 60, 180, 300.
  Afamelanotide: 16mg subcutaneous implant. Placebo: Placebo subcutaneous implant.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 49 | 51
Completed | 47 | 46
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Customized [Mean (Standard Deviation); unit: years] — Between 18-70 years.
  years
    Age | 38.5 (13.3) | 39.2 (12.4) | 38.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 19 | 28 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 49 | 50 | 99
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Days of Phototoxic Reactions (Study Efficacy Population)
Description: The cumulative number of days where a phototoxic reaction occurred was recorded in the patient diary. The reported data represent a cumulative total for days of phototoxic reactions.
  The participant scored the level of pain using an 11-point Likert pain scale, with minimum of 0 and maximum of 10. The 11-point Likert Pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
  The primary analysis population for efficacy was revised, to analyze only participants who reported cumulative total Likert pain scores of at least 26 during the study (0-360 days). This population, which was comprised of 60 patients, is identified as the Efficacy population. Participants with less than 26 Likert pain scores were not included in the analysis.
Time Frame: 0-360 days or Early Termination
Population: Participants who reported a cumulative total Likert pain score of at least 26 during the study (0-360 days), which was comprised of 60 patients, is identified as the Efficacy population.
Measure: Number; unit: Days
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 60 | 60
Days
  Severe Pain | 39 | 45
  Moderate Pain | 129 | 179
  Mild Pain | 1126 | 1237
  No Pain | 8650 | 8484

2. Primary Outcome: The Mean Number of Phototoxic Reactions (Study Efficacy Population)
Description: The mean number of phototoxic reactions that occurred whilst patients were on active compared with placebo implants.
  The days on which the participant experienced pain as a result of phototoxic reactions (caused by exposure to natural light) was recorded in a study diary. On each day such a reaction occurred, the participant scored the level of pain using an 11-point Likert pain scale, with minimum of 0 and maximum of 10. The 11-point Likert pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
  The primary analysis population for efficacy was revised, to analyze only participants who reported a cumulative total Likert pain score of at least 26 during the study (0-360 days). This population, which was comprised of 60 patients, is identified as the Efficacy population.
  Participants with less than 26 Likert pain scores were not included in the analysis.
Time Frame: 0-360 days or Early Termination
Population: The result is reported in a "per sequence" format with the different time points at which the interventions were switched.
  Total of 60 Participants: 32 participants in Group A and 28 participants in Group B.
Measure: Mean (Standard Deviation); unit: counts of episodes
Groups:
- Group A: Afamelanotide: 16mg subcutaneous implant
  Of the 60 participants, 32 were in treatment Group A (active implants on Days 0, 120, 240 and placebo implants on Days 60, 180, 300) and 28 in treatment Group B (placebo implants on Days 0, 120, 240 and active implants on Days 60, 180, 300).
- Group B: Placebo: Placebo subcutaneous implant.
  Of the 60 participants, 32 were in treatment Group A (active implants on Days 0, 120, 240 and placebo implants on Days 60, 180, 300) and 28 in treatment Group B (placebo implants on Days 0, 120, 240 and active implants on Days 60, 180, 300).
Arm/Group | Group A | Group B
Number analyzed (Participants) | 32 | 28
counts of episodes
  Day 0 | 1.44 (3.25) | 2.64 (5.33)
  Day 60 | 0.56 (1.87) | 0.11 (0.31)
  Day 120 | 1.09 (2.08) | 0.79 (2.25)
  Day 180 | 0.32 (2.07) | 0.78 (0.61)
  Day 240 | 0.63 (1.52) | 2.21 (3.57)
  Day 300 | 0.72 (1.42) | 1.96 (4.53)

3. Secondary Outcome: Cumulative Number of Days With Sunlight Exposure (Study Efficacy Population)
Description: The number of days with sunlight exposure was recorded in the patient diary. The sunlight exposures were divided into the following categories: none, < 1 hour, 1 to 3 hours, 3 to 6 hours and > 6 hours per day.
Time Frame: 0-360 days or Early Termination
Population: The primary analysis population for efficacy was revised, with an additional criterion of a total cumulative pain score of at least 26, and omitting patients who did not complete the study. This population, which was comprised of 60 patients, is identified as the Efficacy population.
Measure: Number; unit: Days
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 60 | 60
Days
  > 6 hrs per day | 339 | 250
  3 - 6 hrs per day | 969 | 854
  1 - 3 hrs per day | 2810 | 2695
  < 1 hr per day | 1468 | 1564
  None per day | 4358 | 4582

4. Secondary Outcome: Skin Melanin Density (Study Completers Population)
Description: Changes in melanin density (MD) (measured by spectrophotometry) at each visit by group.
  Participants had their skin pigmentation measured by a non-invasive quantitative skin chromaticity (reflectance) reading. Reflectance by the skin of light measured at the wavelengths of 400 nm and 420 nm was recorded using a Minolta cm-2500d spectrophotometer at the following skin sites: forehead, left cheek, right inside upper arm, left medial forearm, right side of abdomen (avoiding implant insertion site), left side of sacral region/buttock.
  Melanin density was determined for each skin site using the method of Dwyer et al 1998.
Time Frame: Day0, Day14, Day30, Day60, Day74, Day90, Day120, Day150, Day180, Day210, Day240, Day270, Day300, Day330, Day360 or Early Termination
Population: The secondary analysis population for efficacy included those subjects who received all required doses of investigational product. This population is identified as the study completers population.
  Calculated MD <0 or >6 were omitted.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Group A | Group B
Number analyzed (Participants) | 49 | 51
unitless
  Day 0: number analyzed (Participants) | 46 | 46
  Day 0 | 3.42 (0.83) | 3.22 (1.01)
  Day 14: number analyzed (Participants) | 48 | 47
  Day 14 | 3.75 (0.77) | 3.39 (0.95)
  Day 30: number analyzed (Participants) | 47 | 46
  Day 30 | 3.86 (0.72) | 3.40 (1.01)
  Day 60: number analyzed (Participants) | 46 | 46
  Day 60 | 3.80 (0.77) | 3.34 (1.00)
  Day 74: number analyzed (Participants) | 46 | 46
  Day 74 | 3.70 (0.85) | 3.71 (0.89)
  Day 90: number analyzed (Participants) | 46 | 46
  Day 90 | 3.67 (0.80) | 3.75 (0.87)
  Day 120: number analyzed (Participants) | 47 | 46
  Day 120 | 3.52 (0.79) | 3.71 (0.83)
  Day 150: number analyzed (Participants) | 47 | 45
  Day 150 | 3.79 (0.82) | 3.57 (0.89)
  Day 180: number analyzed (Participants) | 47 | 46
  Day 180 | 3.84 (0.74) | 3.50 (0.89)
  Day 210: number analyzed (Participants) | 45 | 46
  Day 210 | 3.76 (0.76) | 3.93 (0.75)
  Day 240: number analyzed (Participants) | 47 | 46
  Day 240 | 3.68 (0.81) | 3.89 (0.73)
  Day 270: number analyzed (Participants) | 43 | 43
  Day 270 | 3.97 (0.72) | 3.81 (0.72)
  Day 300: number analyzed (Participants) | 43 | 43
  Day 300 | 3.89 (0.72) | 3.76 (0.72)
  Day 330: number analyzed (Participants) | 45 | 42
  Day 330 | 3.82 (0.73) | 4.08 (0.63)
  Day 360: number analyzed (Participants) | 42 | 40
  Day 360 | 3.73 (0.69) | 3.97 (0.69)

5. Secondary Outcome: Change in Quality of Life Using SF36 Questionnaire (Physical Component Score) for Study Completers Population
Description: The Summary of SF36 change from Baseline of Physical Component Score (PCS) to the scores during treatment on Days 60, 120, 180, 240, 300 and 360 using the SF36 questionnaire.
  The SF-36 (The Short Form 36 Health Survey) consists of eight scaled scores, which are the weighted sums of the questions in each section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.
  The higher scores represent better health-related quality-of-life.
Time Frame: Day0, Day60, Day120, Day180, Day240, Day300, Day360 or Early Termination
Population: The secondary analysis population for efficacy included those subjects who received all required doses of investigational product. This population, which was comprised of 93 patients, is identified as the study completers population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 47 | 46
score on a scale
  Day 0 | 51.90 (7.05) | 54.22 (5.48)
  Day 60: number analyzed (Participants) | 47 | 45
  Day 60 | 54.20 (5.99) | 54.85 (5.59)
  Day 120 | 54.26 (5.53) | 54.68 (5.78)
  Day 180 | 53.39 (5.88) | 53.72 (5.59)
  Day 240 | 53.19 (7.09) | 54.25 (5.22)
  Day 300 | 53.48 (5.71) | 53.88 (4.93)
  Day 360: number analyzed (Participants) | 47 | 45
  Day 360 | 52.30 (6.03) | 54.88 (5.01)

6. Secondary Outcome: Change in Quality of Life Using SF36 Questionnaire (Mental Component Score) for Study Completers Population
Description: The Summary of SF36 change from Baseline of Mental Component Score (MCS) to the scores during treatment on Days 60, 120, 180, 240, 300 and 360 using the SF36 questionnaire.
  The SF-36 (The Short Form 36 Health Survey) consists of eight scaled scores, which are the weighted sums of the questions in each section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight.
  The higher scores represent better health-related quality-of-life.
Time Frame: Day0, Day60, Day120, Day180, Day240, Day300, Day360 or Early Termination
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A | Group B
Number analyzed (Participants) | 47 | 46
score on a scale
  Day 0 | 51.41 (6.61) | 53.03 (6.75)
  Day 60: number analyzed (Participants) | 47 | 45
  Day 60 | 52.31 (9.58) | 52.26 (7.46)
  Day 120 | 53.16 (7.34) | 52.71 (7.39)
  Day 180 | 53.84 (7.12) | 52.06 (7.50)
  Day 240 | 51.96 (8.48) | 52.34 (8.07)
  Day 300 | 52.99 (9.21) | 52.76 (7.61)
  Day 360: number analyzed (Participants) | 47 | 45
  Day 360 | 52.44 (8.13) | 52.23 (8.00)

ADVERSE EVENTS:
Time Frame: Day 1 - Day 360 or Early Termination
Arm/Group | Afamelanotide | Placebo
Serious Adverse Events (participants affected / at risk) | 3/100 | 3/100
Other Adverse Events (participants affected / at risk) | 94/100 | 88/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=100) | Placebo (N=100)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=100) | Placebo (N=100)
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 13 | 13
Nausea (Gastrointestinal disorders) | 34 | 19
Toothache (Gastrointestinal disorders) | 4 | 7
Vomiting (Gastrointestinal disorders) | 8 | 6
Fatigue (General disorders) | 12 | 11
Implant site haematoma (General disorders) | 8 | 8
Implant site pain (General disorders) | 8 | 6
Oedema peripheral (General disorders) | 5 | 2
Pyrexia (General disorders) | 7 | 4
Influenza (Infections and infestations) | 13 | 4
Nasopharyngitis (Infections and infestations) | 17 | 16
Upper respiratory tract infection (Infections and infestations) | 7 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Dizziness (Nervous system disorders) | 12 | 5
Headache (Nervous system disorders) | 45 | 38
Migraine (Nervous system disorders) | 7 | 8
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Flushing (Vascular disorders) | 8 | 0
Haematoma (Vascular disorders) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No